CLINICAL TRIAL: NCT05473234
Title: Azithromycin for Severe Acute Malnutrition in CMAM, Nigeria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was halted due to low follow-up rates and issues with data collection
Sponsor: University of California, San Francisco (Other)
Collaborators: The Taimaka Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-36912
Record Dates: First submitted 2022-07-11; First posted 2022-07-25 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Experimental): Children in this arm will receive one dose of amoxicillin.
  Interventions: Drug: Azithromycin
- Amoxicillin (Active Comparator): Children in this arm will receive a 5-day course of amoxicillin (standard care).
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Azithromycin — Children enrolled in the trial and randomized to receive azithromycin will receive a single dose of azithromycin at 20 mg/kg up to the maximum adult dose of 1g. Oral azithromycin will be administered at the time of enrollment. Enrolled children will also receive RUTF.
  Arms: Azithromycin
Drug: Amoxicillin — Children enrolled in the trial and randomized to receive amoxicillin will receive a 5-day course of amoxicillin to be given in twice-daily doses of 15 mg/kg per the Nigeria guidelines for severe acute malnutrition. The first dose will be administered at the time of enrollment, and the remaining doses will be administered by the caregiver at home. Enrolled children will also receive RUTF.
  Arms: Amoxicillin

SUMMARY:
This randomized controlled trial is designed to determine the effect of administration of azithromycin compared to amoxicillin as part of the treatment of uncomplicated severe acute malnutrition (SAM) in children aged 6-59 months on weight gain and nutritional recovery. The investigators will randomize children presenting to Taimaka-run nutritional programs at health centers in Gombe State, Nigeria to a single dose of oral azithromycin or a short course of oral amoxicillin upon admission into the program. Apart from the administration of antibiotics, all children will receive standard outpatient treatment for uncomplicated SAM as specified in the guidelines of the government of Nigeria, which includes therapeutic feeding with ready-to-use therapeutic food (RUTF). Enrolled children will be followed weekly at each routine clinic follow-up visit up until nutritional recovery. All enrolled children will return for a final study visit at 8 weeks following enrollment. Anthropometric and vital status data will be collected at each follow-up visit. Weight gain and nutritional recovery over the 8-week study period will be compared by arm as a primary outcome and at 12 weeks as a secondary outcome.

ELIGIBILITY:
Inclusion criteria (all must be met):

* Age 6-59 months
* Weight-for-height z-score (WHZ) < -3 SD or mid-upper arm circumference (MUAC) < 115 mm
* No nutritional or nutritional edema Grade I and II
* Primary residence within catchment area of enrollment site
* Available for full 8-week study
* Has not been admitted to a nutritional program for the treatment of severe acute malnutrition (SAM) in the 2 preceding weeks
* No antibiotic use in past 7 days
* No clinical complications requiring antibiotic treatment
* No clinical complications requiring inpatient treatment
* No congenital abnormality or chronic debilitating illness that would lead to predictable growth faltering or reduce likelihood of SAM treatment benefit (such as cerebral palsy, Down syndrome, congenital heart disease, cleft lip/palate, sickle cell disease, etc)
* No allergy to macrolides/azalides
* Sufficient appetite according to a feeding test with ready-to-use therapeutic food (RUTF)
* Appropriate written informed consent from at least one parent or guardian

Exclusion criteria (any excludes):

* Age < 6 months or > 59 months
* WHZ ≥ -3 SD or MUAC ≥ 115 mm
* Primary residence outside catchment area of enrollment site
* Not available for full 8-week study
* Presence of nutritional edema Grade III
* Admission to a nutritional program for the treatment of SAM in the 2 preceding weeks
* Antibiotic use in past 7 days
* Clinical complications requiring antibiotic treatment
* Clinical complications requiring inpatient treatment
* Congenital abnormality or chronic debilitating illness that would lead to predictable growth faltering or reduce likelihood of SAM treatment benefit (such as cerebral palsy, Down syndrome, congenital heart disease, cleft lip/palate, etc)
* Allergy to macrolides/azalides
* Insufficient appetite according to a feeding test with ready-to-use therapeutic food (RUTF)
* Parent or guardian refuses to provide consent

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieran S O'Brien, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- The Tamaika Project, Gombe, Gombe State, Nigeria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amoxicillin | Azithromycin
Started | 151 | 159
8 Weeks | 96 | 120
Completed (12 weeks) | 42 | 58
Not Completed | 109 | 101

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin | Azithromycin | Total
Number analyzed (Participants) | 151 | 159 | 310
Age, Continuous [Mean (Standard Deviation); unit: month] | 15.79 (7.8) | 16.52 (8.7) | 16.16 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 157
  Male | 75 | 78 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 151 | 159 | 310
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Nigeria | 151 | 159 | 310

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain at 8 Weeks
Description: Weight will be measured at baseline and weekly follow ups, and weight gain will be calculated at 8 weeks in g/day
Time Frame: 8 weeks
Population: 96 children in Amoxicillin arm and 120 children in Azithromycin arm had anthropometry form collected between the 8 weeks window (42 to 70 days)
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 96 | 120
g/day | 30.42 (17.11) | 27.75 (18.82)

2. Secondary Outcome: Number of Participants With Nutritional Recovery at 8 Weeks
Description: Nutritional recovery will be defined as a child having WHZ ≥ -2 on two consecutive visits and no acute complication or edema for the past 7 days AND / OR MUAC of ≥ 125mm on 2 consecutive visits and no acute complication or edema for the past 7 days.
  Children will be considered recovered or not recovered using these criteria
  Anthropomorphic outcomes are defined according to the World Health Organization's 2006 Child Growth Standards
  A z-score of 0 represents the population median. The z-score will be positive if the data value lies above the mean, and it will be negative if the value lies below the median. A WHZ < -2 standard distributions below the median is defined as moderately wasted, while a WHZ < -3 standard distributions below the median is defined as severely wasted.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 96 | 120
Participants | 85 | 105

3. Other Pre Specified Outcome: Weight Gain Over 12 Weeks
Description: Weight will be measured at baseline and weekly follow up visits for 8 weeks, and at 12 weeks after admission to the program. Weight gain will be defined as grams per kilogram per day (g/day).
Time Frame: 12 weeks
Population: 42 children in Amoxicillin arm and 58 children in Azithromycin arm had anthropometry form collected between the 12 weeks window (70 to 98 days)
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
g/day | 22.67 (13.13) | 23.89 (11.58)

4. Other Pre Specified Outcome: Time to Recovery
Description: Time from enrollment to nutritional recovery will be calculated in days by subtracting the date of enrollment from the date of nutritional recovery.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 133 | 150
days | 21.4 (19.2) | 22.4 (19.3)

5. Other Pre Specified Outcome: Nonresponse at 8 Weeks
Description: Number of children with nonresponse will be documented if a child does not meet the criteria for nutritional recovery at 8 weeks after enrollment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 96 | 120
Participants | 11 | 15

6. Other Pre Specified Outcome: Number of Participants Who Transferred to Inpatient Care
Description: The occurrence, date, and reason for transfer from outpatient to inpatient treatment will be recorded.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
Participants | 3 | 4

7. Other Pre Specified Outcome: Mortality by 8 Weeks
Description: Vital status will be assessed at baseline and at weekly follow up visits for 8 weeks, and mortality will be defined as death during the study period. Date of death will be recorded.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 96 | 120
Participants | 3 | 2

8. Other Pre Specified Outcome: Mortality by 12 Weeks
Description: Vital status will be assessed at baseline, weekly follow up visits for 8 weeks, and at 12 weeks, and mortality will be defined as death during the study period. Date of death will be recorded.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
Participants | 4 | 3

9. Other Pre Specified Outcome: Clinical Signs of Infection
Description: Number of participants with clinical sign of infection will be recorded At baseline, weekly follow up visits for 8 weeks, and at the 12-week follow up visit, including care-giver reported experience of fever, diarrhea, vomiting, and respiratory infection/cough and clinical diagnoses made at by site personnel
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 32 | 50
Participants | 6 | 16

10. Other Pre Specified Outcome: Height-for-age Z-score (HAZ)
Description: Height or length will be measured monthly (baseline and the 4-, 8-, and 12-week follow up visits) and height-for-age z-scores will be calculated.
  Anthropomorphic outcomes are defined according to the World Health Organization's 2006 Child Growth Standards
  A z-score of 0 represents the population median. The z-score will be positive if the data value lies above the mean, and it will be negative if the value lies below the median. A HAZ < -2 standard distributions below the median is defined as stunted, while a HAZ < -3 standard distributions below the median is defined as severely stunted.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
z score | -3.77 (1.98) | -3.64 (1.49)

11. Other Pre Specified Outcome: Mid-upper Arm Circumference (MUAC)
Description: Mid-upper arm circumference (centimeters) will be measured at all follow-up time points (baseline, weekly follow up visits for 8 weeks, and at the 12-week follow up visit).
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
centimeters (cm) | 12.70 (0.70) | 12.73 (0.52)

12. Other Pre Specified Outcome: Weight-for-age Z-score (WAZ)
Description: Weight will be measured at all follow-up time points (baseline, weekly follow up visits for 8 weeks, and at the 12-week follow up visit) and weight-for-age z-scores will be calculated.
  Anthropomorphic outcomes are defined according to the World Health Organization's 2006 Child Growth Standards
  A z-score of 0 represents the population median. The z-score will be positive if the data value lies above the mean, and it will be negative if the value lies below the median. A WAZ < -2 standard distributions below the median is defined as underweight, while a WAZ < -3 standard distributions below the median is defined as severely underweight.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
z score | -2.67 (1.31) | -2.48 (0.95)

13. Other Pre Specified Outcome: Weight-for-height Z-score (WHZ)
Description: Weight and height, assessed at all follow-up time points (baseline, weekly follow up visits for 8 weeks, and at the 12-week follow up visit), will be used to calculate weight-for-height z-scores.
  Anthropomorphic outcomes are defined according to the World Health Organization's 2006 Child Growth Standards
  A z-score of 0 represents the population median. The z-score will be positive if the data value lies above the mean, and it will be negative if the value lies below the median. A WHZ < -2 standard distributions below the median is defined as moderately wasted, while a WAZ < -3 standard distributions below the median is defined as severely wasted.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 42 | 58
z score | -0.69 (1.44) | -0.60 (1.54)

14. Other Pre Specified Outcome: Malaria
Description: Rapid diagnostic tests for malaria will be conducted at baseline and week 8 to determine malaria infection status. Positivity rate will be compared between arms
Time Frame: 8 weeks
Population: 55 children in Amoxicillin arm and 66 children in Azithromycin arm had malaria test between the 8 weeks window (42 to 70 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin | Azithromycin
Number analyzed (Participants) | 55 | 66
Participants | 9 | 16

ADVERSE EVENTS:
Time Frame: Parents or guardians of enrolled children will be instructed to report any adverse events experienced within the 7 days following the enrollment visit, by phone or in person. All cause-mortality will be monitored until 12 weeks.
Description: Parents or guardians of enrolled children were instructed to report any adverse events experienced within the 7 days following the enrollment visit, by phone or in person. There were 133 participants in Amoxicillin arm and 142 participants in Azithromycin arm had follow-ups at 7 days.
  All cause-mortality was monitored until 12 weeks. There were 42 participants in Amoxicillin arm and 58 participants in Azithromycin arm had follow-ups at 12 weeks.
Arm/Group | Amoxicillin | Azithromycin
All-Cause Mortality (participants affected / at risk) | 4/42 | 3/58
Serious Adverse Events (participants affected / at risk) | 1/133 | 0/142
Other Adverse Events (participants affected / at risk) | 1/133 | 3/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amoxicillin (N=133) | Azithromycin (N=142)
Death in 7 days (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amoxicillin (N=133) | Azithromycin (N=142)
weight loss (General disorders) | 1 | 1
severe fever (General disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05473234/Prot_SAP_000.pdf